CLINICAL TRIAL: NCT05860894
Title: Post Intensive Care Unit Atrial Fibrillation
Acronym: PIAF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A01292-41
Record Dates: First submitted 2023-01-27; First posted 2023-05-16 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation; Critical Illness
Keywords: intensive care unit; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implantable ECG holter device (Experimental): Adult patients with new onset atrial fibrillation occuring in the ICU will be implanted with an implantable ECG holter device (Biomonitor3, Biotronik) to monitor arrhythmia episodes up to 2 years after ICU discharge.
  Interventions: Device: Implantable ECG holter device (Biomonitor3, Biotronik)

INTERVENTIONS:
Device: Implantable ECG holter device (Biomonitor3, Biotronik) — Subcutaneous implantation of ECG holder device to monitor ECG

SUMMARY:
Atrial fibrillation (AF) is a common heart rhythm disorder in the intensive care unit (ICU). It can be precipitated by multiple factors but it is unclear whether AF persists after discharge from the ICU, and long term. This study will investigate whether AF recurs up to one year after ICU discharge.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common heart rhythm disorder encountered in the intensive care unit (ICU). It can be precipitated by multiple factors present in critically ill patients, such as tissue hypoxia, metabolic disorders etc. There is a paucity of data regarding the persistence of AF in these patients after discharge from the ICU, and in the longer term. Therefore, this study will investigate whether AF recurs up to one year after ICU discharge using an implantable ECG Holter device in adult patients discharged alive from the ICU, with documented new onset AF.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* New onset atrial fibrillation diagnosed in the ICU (12 lead ECG or documented episode of atrial fibrillation lasting at least 30 seconds)
* Patient hospitalized in the ICU with at least one of the following two criteria:

  * orotracheal intubation for mechanical ventilation
  * AND/OR treatment with amines (vasopressors or inotropic agents)
* Written informed consent
* Patient affiliated to a social security regime (or beneficiary thereof)

Exclusion Criteria:

* Documented history of atrial fibrillation
* patients admitted to the ICU after cardiothoracic surgery
* Patients with life expectancy <12 months
* Patients under legal or judicial protection
* Patients with no social security coverage
* Patients within the exclusion period of another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrence of atrial fibrillation | up to 1 year after ICU discharge
  Any episode of atrial fibrillation, atrial tachycardia or atrial flutter lasting at least 1 minute, as documented on the implantable device recordings

SECONDARY OUTCOMES:
Burden of atrial fibrillation in absolute value | up to 2 years after ICU discharge
  Burden of atrial fibrillation assessed as time (in days, hours and minutes), expressed as a absolute value
Burden of atrial fibrillation (percentage of time spent in atrial fibrillation) | up to 2 years after ICU discharge
  Burden of atrial fibrillation assessed as time (in days, hours and minutes) expressed as a percentage time spent in atrial fibrillation
Rate of Stroke | up to 2 years after ICU discharge
  Ischemic or hemorrhagei stroke documented by imaging, major bleeding (ISTH classification) or documented peripheral emboli
Number of participants with Change in treatment | up to 2 years after ICU discharge
  Changes in treatment due to the discovery of atrial fibrillation

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No